CLINICAL TRIAL: NCT06429085
Title: Rex Robot Assisted Rehabilitation to Enhance Balance and Mobility for People With Multiple Sclerosis, Clinical and Biomarker Study - RAPPER IV
Acronym: RAPPER IV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: East Kent Hospitals University NHS Foundation Trust (Other Government)
Collaborators: Rex Bionics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol Version 2.0
Record Dates: First submitted 2024-05-13; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
Keywords: Balance; Core stability; Mobility; Powered exoskeleton; Neuro-rehabilitation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Prospective, open label, single arm, non-randomized, non-comparative feasibility study of Rex robot assisted training to improve balance and mobility for people living with MS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- People diagnosed with Multiple Sclerosis (Experimental): Use of powered Rex robotic exoskeleton to enable the practice of core stability balance exercises
  Interventions: Device: Rex robotic assisted balance exercises

INTERVENTIONS:
Device: Rex robotic assisted balance exercises — Individual is supported by a Rex robotic exoskeleton which enables assisted and supervised practise of balance exercises. This intervention took place as a supported and supervised series of 5 sessions over 5 weeks as an Out-patient.

SUMMARY:
Multiple Sclerosis (MS) poses challenges to balance and mobility, impacting the daily lives of affected individuals. The RAPPER IV study is a clinical trial to evaluate a balance and mobility training intervention supported by a powered Rex robotic exoskeleton for people living with MS.

Aims and objectives:

This study aims to gain an insight into the potential health benefits of using a Rex robot to assist in a neuro-rehabilitation intervention program focused on improving balance and functional mobility with supervision from a specialist clinician.

Objectives

* to evaluate the feasibility of using the Rex robotic walking device for rehabilitation with people who have mobility restrictions due to Multiple Sclerosis (MS)
* to assess and evaluate the clinical effectiveness of a 5-week robotic assisted exercise program focused on core stability exercises, balance and walking using patient related outcome measures
* to gain an insight into the experiences of participants and their spouses of using the robotic walking device for rehabilitation and how this has impacted on their lives

A single cohort group of 20 people who were living with MS who met trial eligibility criteria were recruited. A variety of clinical outcome measurements were taken pre, during and post trial and results were analysed by a statistician.

DETAILED DESCRIPTION:
The key research questions:

* Is it feasible for a person with balance and mobility impairment caused by MS to use a robotic walking device to exercise in standing and walking with supervision safely?
* What are the key outcome measures most sensitive to measurable change in this study population sample, which may reflect potential improvement during the trial period? (Clinical outcome scales and self-reported questionnaires)
* Is this robotic assisted balance and mobility training program feasible, safe and effective?
* Does the completion of this balance and mobility exercise treatment intervention result in measurable improvements in balance, mobility, spasticity, lower limb joint range of movement and achievable individual patient goals?

To answer these questions, we invited 20 people diagnosed with MS (as defined by "McDonald" criteria, Polman et al, 2011) to undertake a 5-week balance exercise intervention program supported by the use of the Rex robotic walking device, designed to strengthen their postural body and leg muscles and improve their balance.

Participants were monitored and progressed on an individual basis throughout the treatment program as appropriate and a range of standardised assessments, questionnaires and relevant clinical outcome scales were used to capture and measure change related to this trial.

Prospective, open label, single arm, non-randomized, non-comparative feasibility study of Rex robot assisted training to improve balance, mobility and cardiovascular fitness for people living with MS.

A purposive sample of 20 adults, who have a primary diagnosis of MS, aged between 18 and 80 years old, with an Expanded Disability Status Scale (EDSS) as defined by Kurtzke (1983), with scores between 4 and 6.5 were recruited into this study.

ELIGIBILITY:
Inclusion Criteria:

* • Are aged greater than 18 years and less than 80 years

  * Have a confirmed diagnosis of MS by a Consultant Neurologist as per McDonald Criteria.
  * Have moderate mobility restriction as defined by an Extended Disability Status Scale (EDSS) score of between 4 to 6.5
  * Ten participants to be recruited from EDSS 4 to 5.5
  * Ten participants to be recruited from EDSS 5.5 to 6.5
  * Within the anthropometric requirements of the REX device (See 'RAPPER III- MS 014 TF-04 v 3.0 REX Clinical Assessment Guide A4' for details of weight, height, size and range of motion requirements)
  * Offer written informed consent to take part in the study

Exclusion Criteria:

* a history of osteoporosis or osteoporosis related bone fractures.
* skin integrity issues that could be adversely affected by the REX device
* severe hypertonia (spasticity) as indicated by a score equal to or greater than 4 on the modified Ashworth scale for any muscle in their lower limbs.
* a behavioural, cognitive or communication impairment which could interfere with the ability to participate in a rehabilitation program, as noted during screening (e.g., agitation, inability to follow two step commands)
* are unable or unwilling to provide informed consent
* are considered medically unsuitable for rehabilitation in the opinion of the screening medical specialist
* a known allergy (skin contact) to materials used in Rex
* are pregnant
* taking part in any other medical research trial at the same time

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Timed transfer into the Rex device | Time point 1 - Week 1
  Timed transfer into the Rex device with appropriate level of assistance
Completion of sit to stand and stand to sit within the Rex device | Time point 1 - Week 1
  Completion of sit to stand and stand to sit within the Rex device with hands on assistance from trial therapist
Completion of 1 Rex robotic assisted balance rehabilitation exercise session | Time point 1 - Week 1
  Completion of 1 Rex robotic assisted balance rehabilitation exercise session with hands on assistance from trial therapist
Screening loss analysis | End of recruitment period - Week 30
  Number of individuals screened and those eligible who entered the trial and those who completed the trial

SECONDARY OUTCOMES:
Timed up and Go | Time point 1 - Week 1
  Timed up and Go
Berg Balance Scale | Measured at 3 time points: Weeks 1, 6 and 10
  Berg Balance Scale
Visual Analog Scale (Pain) | Measured at 2 time points: Weeks 1 and 6
  Visual Analog Scale (Pain)
Modified Falls Efficacy Scale | Measured at 2 time points: Weeks 1 and 6
  Balance and falls risk
Activities-specific Balance Confidence scale | Measured at 2 time points: Weeks 1 and 6
  Balance and confidence in balance
Spasticity Impact Scale | Measured at 2 time points: Weeks 1 and 6
  Perception of impact of spasticity on life
EQ-5D-5L | Measured at 2 time points: Weeks 1 and 6
  Perceived Health Related Quality of Life
MSIS-29 | Measured at 2 time points: Weeks 1 and 6
  Perceived impact of MS on life
Joint range of movement | Measured at 2 time points: Weeks 1 and 6
  Joint range of movement
Goal Attainment Scale | Set at Week 1 and measured and reviewed at Week 25
  Goal Attainment Scale
Modified Ashworth Scale | Measured at 2 time points: Weeks 1 and 6
  Modified Ashworth Scale for muscle spasticity

CONTACTS AND LOCATIONS:
Locations (1):
- East Kent Hospitals University NHS Trust, Canterbury, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zajicek J, Fox P, Sanders H, Wright D, Vickery J, Nunn A, Thompson A; UK MS Research Group. Cannabinoids for treatment of spasticity and other symptoms related to multiple sclerosis (CAMS study): multicentre randomised placebo-controlled trial. Lancet. 2003 Nov 8;362(9395):1517-26. doi: 10.1016/S0140-6736(03)14738-1. PMID 14615106
- [Result] Straudi S, Fanciullacci C, Martinuzzi C, Pavarelli C, Rossi B, Chisari C, Basaglia N. The effects of robot-assisted gait training in progressive multiple sclerosis: A randomized controlled trial. Mult Scler. 2016 Mar;22(3):373-84. doi: 10.1177/1352458515620933. Epub 2015 Dec 10. PMID 26658817
- [Result] Bethoux F, Bennett S. Introduction: enhancing mobility in multiple sclerosis. Int J MS Care. 2011 Spring;13(1):1-3. doi: 10.7224/1537-2073-13.1.1. No abstract available. PMID 24453699
- [Result] Latimer-Cheung AE, Pilutti LA, Hicks AL, Martin Ginis KA, Fenuta AM, MacKibbon KA, Motl RW. Effects of exercise training on fitness, mobility, fatigue, and health-related quality of life among adults with multiple sclerosis: a systematic review to inform guideline development. Arch Phys Med Rehabil. 2013 Sep;94(9):1800-1828.e3. doi: 10.1016/j.apmr.2013.04.020. Epub 2013 May 10. PMID 23669008
- [Result] Donze C. Update on rehabilitation in multiple sclerosis. Presse Med. 2015 Apr;44(4 Pt 2):e169-76. doi: 10.1016/j.lpm.2014.10.019. Epub 2015 Mar 4. PMID 25746432
- [Result] Wiles CM, Newcombe RG, Fuller KJ, Shaw S, Furnival-Doran J, Pickersgill TP, Morgan A. Controlled randomised crossover trial of the effects of physiotherapy on mobility in chronic multiple sclerosis. J Neurol Neurosurg Psychiatry. 2001 Feb;70(2):174-9. doi: 10.1136/jnnp.70.2.174. PMID 11160464
- [Result] Cattaneo D, Jonsdottir J, Zocchi M, Regola A. Effects of balance exercises on people with multiple sclerosis: a pilot study. Clin Rehabil. 2007 Sep;21(9):771-81. doi: 10.1177/0269215507077602. PMID 17875557
- [Result] Birch N, Graham J, Priestley T, Heywood C, Sakel M, Gall A, Nunn A, Signal N. Results of the first interim analysis of the RAPPER II trial in patients with spinal cord injury: ambulation and functional exercise programs in the REX powered walking aid. J Neuroeng Rehabil. 2017 Jun 19;14(1):60. doi: 10.1186/s12984-017-0274-6. PMID 28629390
- [Result] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Result] Sakel M, Saunders K, Hodgson P, Stephensen D, Phadke CP, Bassett PA, Wilkinson D. Feasibility and Safety of a Powered Exoskeleton for Balance Training for People Living with Multiple Sclerosis: A Single-Group Preliminary Study (Rapper III). J Rehabil Med. 2022 Dec 9;54:jrm00357. doi: 10.2340/jrm.v54.4544. PMID 36484722